CLINICAL TRIAL: NCT01571830
Title: Improving Nutrient Intake and Growth in Children With Multiple Food Allergies
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Other Study IDs: CHW 11/181, GC 1404
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Food Allergy
Keywords: food allergy; nutrient intake; growth
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
* Hypothesis 1: Food allergies are associated with poor growth which can be corrected with nutrition intervention.

  * More than 10% of children with multiple food allergies will have a weight-for-age z-score less than - 2 at diagnosis. The z-score is a measure of the distance from the mean value, or 50th percentile on the growth chart. A z-score of less than - 2 indicates that the child is underweight.
  * Growth parameters of children with multiple food allergies will improve after intervention by a team that includes a dietitian and an allergist.
* Hypothesis 2: Food allergies are associated with low micronutrient intake which can be corrected with nutrition intervention.

  o More than 30% of children with multiple food allergies will consume less than 67% of the Dietary Reference Intake for at least one macronutrient or micronutrient at diagnosis.
* Macronutrient and micronutrient intake will increase after intervention by a team that includes a dietitian and an allergist.

o

• Hypothesis 3: Food allergies are related to behavioral feeding problems which can be corrected with nutrition intervention.

* At least 25% of children with multiple food allergies will have behavioral feeding problems at diagnosis.
* Prevalence of behavioral feeding problems will decrease after nutrition intervention.

DETAILED DESCRIPTION:
This is a prospective observational study with repeated measure design. All participants aged 6 months to 6 years diagnosed with two or more food allergies will be invited to participate in the research study. At least one of the two food allergies must be milk, egg, wheat, or soy, which are nutritionally important food allergies. Inclusion criteria include diagnosis of two or more food allergies confirmed with skin prick testing or serum specific IgE (SIgE)testing. Participants aged 12 months or older will be invited to participate in the Mealtime Behavior Questionnaire (MBQ) and Feeding Strategies Questionnaire (FSQ). Participants with developmental delay, genetic syndromes or other chronic medical conditions will be excluded from the study. Participants with two or more food allergies that do not have at least one nutritionally important food allergy (milk, egg, wheat, soy) will not be invited to participate in the study. We will also exclude participants with a history of digestive surgery, non English-speaking patients, and patients currently receiving nutrition support (enteral or parenteral nutrition). Patients will be excluded if they received greater than one week of oral steroids in the previous three months. Exclusively breastfed infants will be excluded from the study as their nutrient intake cannot accurately assessed (must consume at least some foods or formulas). We will include patients if they have asthma, eczema, or both. There will be no control group recruited for the study as comparisons will be made within the study population.

Subjects will be recruited from the Asthma, Allergy, & Immunology Clinic at the main campus of Children's Hospital of Wisconsin. At the first visit with the dietitian, subjects will be enrolled and consent will be obtained. Height, weight, and head circumference (until 2 YO) will be measured and recorded using standard procedures. The Mealtime Behavior Questionnaire (MBQ) and Feeding Strategies Questionnaire (FSQ) will be filled out by the parent or guardian. Demographic data and medical history will be obtained. Height/length, weight, and head circumference from the first allergist visit will be obtained from the medical record and recorded for use in the study. A multiple-pass 24-hour recall will be completed. In addition, they will receive standardized nutrition intervention to include nutrition assessment, food allergy education, and general nutrition education.

The participant will attend a second visit with the dietitian. Height, weight, and head circumference will be measured and recorded using standard procedures. A multiple-pass 24-hour recall will be completed. The participant's parent or guardian will complete the MBQ and FSQ. Follow-up nutrition intervention will include nutrition reassessment, food allergy education as needed, and general nutrition education as needed.

All aspects of this study, with the exception of MBQ, and FSQ, are the current standard of care in the Asthma, Allergy, and Immunology clinic for patients with multiple food allergies.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to 6 years
* 2 or more food allergies
* At least one of the food allergies must be milk, egg, wheat, or soy
* Confirmed with skin prick testing or SIgE
* Diagnosed at CHW Asthma, Allergy, & Immunology Clinic
* Second opinions are included as long as patient has never been seen by a dietitian for food allergies

Exclusion Criteria:

* Previously seen by a dietitian for food allergies
* Developmental delay
* Genetic syndrome
* Other chronic medical conditions besides asthma, eczema, or eosinophilic esophagitis
* Hyper-IgE syndrome
* Immune deficiency disease
* History of digestive surgery
* Non-English speaking
* Currently receiving nutrition support (enteral or parenteral nutrition)
* Received oral steroids for more than 7 days in the previous three months

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: New patients to the Allergy & Immunology outpatient clinic at Children's Hospital of Wisconsin (CHW).
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2011-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Growth | 6 months
  Weight for age, length/height for age, and weight for length/height z-scores will be assessed. Growth will be compared to reference standards. Growth velocity will be calculated in grams/day.

SECONDARY OUTCOMES:
Nutrient intake | 6 months
  Changes in nutrient intake will be assessed using a multiple-pass 24 hour recalls administered at 4 times throughout the 6 month study period. Nutrient intake will be compared with the Dietary Reference Intakes (DRI) and changes in nutrient intake over time will be assessed. The primary goal is to assess changes in nutrient intake before and after nutrition intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Goday, MD, Principal Investigator — Medical College of Wisconsin & Children's Hospital of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Johnson RK, Driscoll P, Goran MI. Comparison of multiple-pass 24-hour recall estimates of energy intake with total energy expenditure determined by the doubly labeled water method in young children. J Am Diet Assoc. 1996 Nov;96(11):1140-4. doi: 10.1016/S0002-8223(96)00293-3. PMID 8906138